CLINICAL TRIAL: NCT00985556
Title: Randomized Phase II Study of S-1 (SOX) or Capecitabine (XELOX) in Combination With Oxaliplatin in Patients With Recurrent or Metastatic Gastric Cancer
Brief Title: Oxaliplatin and S-1 or Oxaliplatin and Capecitabine in Treating Patients With Recurrent, Metastatic, or Unresectable Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000650368; YONSEI-4-2007-0296
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2009-09

CONDITIONS: Gastric Cancer
Keywords: recurrent gastric cancer; adenocarcinoma of the stomach; stage IIIA gastric cancer; stage IIIB gastric cancer; stage IIIC gastric cancer; stage IV gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Oxaliplatin

ARMS (2):
- Arm I (Experimental): Patients receive oral S-1 twice daily on days 1-14 and oxaliplatin IV over 2 hours on day 1.
  Interventions: Drug: oxaliplatin; Drug: tegafur-gimeracil-oteracil potassium
- Arm II (Experimental): Patients receive oral capecitabine twice daily on days 1-14 and oxaliplatin as in arm I.
  Interventions: Drug: capecitabine; Drug: oxaliplatin

INTERVENTIONS:
Drug: capecitabine — Given orally
  Arms: Arm II
Drug: oxaliplatin — Given IV
Drug: tegafur-gimeracil-oteracil potassium — Given orally
  Arms: Arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, S-1, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known whether giving oxaliplatin together with S-1 is more effective than giving oxaliplatin together with capecitabine.

PURPOSE: This randomized phase II trial is studying how well giving oxaliplatin together with S-1 works compared to oxaliplatin given together with capecitabine in treating patients with recurrent, metastatic, or unresectable gastric cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the time to progression in patients with recurrent or metastatic gastric cancer treated with oxaliplatin in combination with S-1 vs capecitabine.

Secondary

* To assess progression-free survival, overall response, disease-control rate, time-to-treatment failure, response duration, time to response, overall survival, safety, quality of life, pharmacogenetics, and psychologic distress/coping strategy.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral S-1 twice daily on days 1-14 and oxaliplatin IV over 2 hours on day 1.
* Arm II: Patients receive oral capecitabine twice daily on days 1-14 and oxaliplatin as in arm I.

Courses in both arms repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the stomach
* Unresectable advanced disease or recurrent disease after resection
* At least one radiographically documented (CT scan or MRI) measurable or evaluable lesion in a previously non-irradiated area according to RECIST
* No clinical evidence of brain metastases or history of other CNS disease unless adequately treated

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Estimated life expectancy > 3 months
* Hemoglobin ≥ 9 g/dL
* White blood cell ≥ 4,000/µL
* ANC ≥ 2,000/µL
* Platelets ≥ 100,000/µL
* Bilirubin ≤ 1.25 times upper limit of normal (ULN) (≤ 2.0 times ULN if hepatic metastasis present)
* Serum creatinine ≤ 1.5 times ULN
* Creatinine clearance ≥ 60 mL/min
* AST/ALT ≤ 3.0 times ULN (≤ 5.0 times ULN if hepatic metastasis present)
* Alkaline phosphatase ≤ 3.0 times ULN (≤ 5.0 times ULN if bone metastasis present)
* Must have an intact gastrointestinal tract
* Able to take oral medications
* No medically uncontrolled severe infections or complications
* No prior malignancy other than gastric cancer in the last 5 years except for basal cell cancer of the skin or preinvasive cancer of the cervix
* Not pregnant or nursing
* No neuropathy ≥ grade 2
* No clinically relevant heart disease
* No evidence of past medical history or psychosocial dysfunction that contraindicates the use of an investigational drug or puts the patient at risk
* No dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent
* No uncontrolled hepatitis B or C, chronic liver disease, or diabetes mellitus
* No other evidence of inappropriate suspicious condition

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for advanced or recurrent disease

  * Prior adjuvant chemotherapy allowed if finished > 6 months before start of study treatment
* No prior therapeutic radiotherapy

  * Prior palliative radiotherapy allowed if it was not done for primary, evaluable, or intraabdominal lesions
* No prior capecitabine or oxaliplatin
* No other concurrent chemotherapy or radiotherapy (except localized radiotherapy for pain relief)
* No concurrent chemically related analogues, such as warfarin, phenytoin, or allopurinol
* No concurrent steroid therapy except as follows:

  * Prophylactic use for hypersensitivity control or antiemetic purpose allowed
  * Chronic low dose of steroid (less than methylprednisolone 20 mg or equivalent dose) allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2009-01

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Hyun C. Chung, MD, PhD, Principal Investigator — Yonsei University
Locations (1):
- Yonsei Cancer Center at Yonsei University Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kang JI, Chung HC, Jeung HC, Kim SJ, An SK, Namkoong K. FKBP5 polymorphisms as vulnerability to anxiety and depression in patients with advanced gastric cancer: a controlled and prospective study. Psychoneuroendocrinology. 2012 Sep;37(9):1569-76. doi: 10.1016/j.psyneuen.2012.02.017. Epub 2012 Mar 28. PMID 22459275